CLINICAL TRIAL: NCT00953927
Title: Phase II Double-blinded Randomized Controlled Evaluation of MVA85A/AERAS-485 for Safety, Immunogenicity and Prevention of Tuberculosis in BCG-vaccinated, HIV-negative Infants
Brief Title: A Study of MVA85A in Healthy Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aeras (Other)
Collaborators: University of Oxford (Other); University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C-020-485; Oxford TB020 (Other: The University of Oxford)
Record Dates: First submitted 2009-07-31; First posted 2009-08-06 (Estimated); Results first posted 2013-12-12 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-04

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — MVA 85A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Investigational Vaccine (Experimental): MVA85A/AERAS-485; subset into cohorts to explore different safety and immunogenicity tests.
  Interventions: Biological: MVA85A/AERAS-485
- Control Group (Placebo Comparator): Candida Skin Test Antigen control; subset into cohorts to explore different safety and immunogenicity tests.
  Interventions: Biological: Candida Skin Test Antigen

INTERVENTIONS:
Biological: MVA85A/AERAS-485 — Attenuated virus MVA vector with insertion. Single dose vaccine, 1 x 10^8 pfu.
  Other Names: Manufactured by IDT of Germany.
  Arms: Investigational Vaccine
Biological: Candida Skin Test Antigen — 1 test, administered once as a placebo control.
  Other Names: Candin(R); Manufactured by Allermed Laboratories of USA.
  Arms: Control Group

SUMMARY:
This was a Phase II double-blinded randomized controlled evaluation of safety, immunogenicity and efficacy of MVA85A/AERAS-485 in Bacillus Calmette-Guérin (BCG) vaccinated infants without tuberculosis or HIV infection. This study planned to enroll 2784 infants (126 to 182 days of age) who received study vaccine or control and were followed for 15 - 36 months. The study was conducted at a single site in South Africa.

DETAILED DESCRIPTION:
This was a Phase II double-blinded randomized controlled evaluation of safety, immunogenicity and efficacy of MVA85A/AERAS-485 in BCG vaccinated infants without tuberculosis or HIV infection. Infants (126 to 182 days) received intradermal (ID) study vaccine (MVA85A/AERAS-485 or Candida skin test antigen control). All infants were to be followed for at least 15 months after the last infant was enrolled into the study. Given completion of enrollment in 21 months, the total duration of follow-up for each infant was scheduled to be at least 15 months and up to 36 months. Infants were to be followed for the entire duration of the study both for the development of tuberculosis and serious adverse events.

On enrollment to the study, eligible infants were assigned to a study group starting with Study Group 1 and were randomized in a 1:1 ratio within a study group to receive either MVA85A/AERAS-485 or Candida skin test antigen control. Infants were assigned to a safety cohort (Study Group 1), then into 1 of 3 immunological assay evaluation groups (Study Groups 2-4), and finally the remainder of infants were assigned into the correlate of protection cohort (Study Group 5). At least 330 infants were to be randomized in Study Group 1, up to 50-60 infants each in Study Groups 2-4, and the remaining infants were randomized in Study Group 5.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 126 through 182 days on the day of randomization (Study Day 0)
2. Written informed consent obtained from the parents/guardian
3. Weight: by chart >3rd percentile on Study Day 0 or, if < 3rd percentile, infant has shown a stable growth pattern
4. BCG vaccination within 7 days of birth
5. Generally good health confirmed by medical history and physical examination within 35 days prior to Study Day 0
6. Must have received age-appropriate doses of pneumococcal vaccine as recommended by the South African Department of Health but no injection within 14 day prior to Study Day 0
7. Ability to complete follow-up period as required by the protocol
8. Completed simultaneous enrollment in the Aeras Vaccine Development Registry protocol

Exclusion Criteria:

1. Acute illness on Study Day 0
2. Fever >=37.5 degrees Celsius on Study Day 0
3. Evidence of significant active infection on Study Day 0
4. Received a Expanded Program of Immunization (EPI) within 14 days prior to Study Day 0
5. Historical or virological evidence of individual or maternal human immunodeficiency virus (HIV-1) infection
6. History of allergic disease or reactions likely to be exacerbated by any component of the study vaccine
7. Previous medical history, or evidence, of an intercurrent illness that may compromise the safety of the infant in the study
8. Evidence of chronic hepatitis from any cause
9. History or evidence of any systemic disease on physical examination or any acute, chronic or intercurrent illness that, in the opinion of the investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine
10. History of or known tuberculosis or treatment for tuberculosis
11. Shared residence since birth with an individual with active tuberculosis or on anti-tuberculosis treatment for less than 2 months

Ages: 126 Days to 182 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2797 (Actual)
Dates: Start 2009-07; Primary Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Tameris, MD, Principal Investigator — South African Tuberculosis Vaccine Initiative; Bernard Landry, MPH, Study Director — Aeras; Helen McShane, MD, Study Chair — University of Oxford; Centre for Vaccinology & Tropical Medicine
Locations (3):
- South Africa (3):
  - South African Tuberculosis Vaccine Initiative (Satellite), Ceres
  - South African Tuberculosis Vaccine Initiative (Satellite), Robertson
  - South African Tuberculosis Vaccine Initiative (Headquarters), Worcester

REFERENCES:
- [Background] Tameris MD, Hatherill M, Landry BS, Scriba TJ, Snowden MA, Lockhart S, Shea JE, McClain JB, Hussey GD, Hanekom WA, Mahomed H, McShane H; MVA85A 020 Trial Study Team. Safety and efficacy of MVA85A, a new tuberculosis vaccine, in infants previously vaccinated with BCG: a randomised, placebo-controlled phase 2b trial. Lancet. 2013 Mar 23;381(9871):1021-8. doi: 10.1016/S0140-6736(13)60177-4. PMID 23391465
- [Background] Tameris M, McShane H, McClain JB, Landry B, Lockhart S, Luabeya AK, Geldenhuys H, Shea J, Hussey G, van der Merwe L, de Kock M, Scriba T, Walker R, Hanekom W, Hatherill M, Mahomed H. Lessons learnt from the first efficacy trial of a new infant tuberculosis vaccine since BCG. Tuberculosis (Edinb). 2013 Mar;93(2):143-9. doi: 10.1016/j.tube.2013.01.003. Epub 2013 Feb 12. PMID 23410889
- [Background] Mulenga H, Tameris MD, Luabeya KK, Geldenhuys H, Scriba TJ, Hussey GD, Mahomed H, Landry BS, Hanekom WA, McShane H, Hatherill M. The Role of Clinical Symptoms in the Diagnosis of Intrathoracic Tuberculosis in Young Children. Pediatr Infect Dis J. 2015 Nov;34(11):1157-62. doi: 10.1097/INF.0000000000000847. PMID 26226446
- [Background] Luabeya KK, Tameris MD, Geldenhuys HD, Mulenga H, Van Schalkwyk A, Hughes EJ, Toefey A, Scriba TJ, Hussey G, Mahomed H, McShane H, Landry B, Hanekom WA, Hatherill M. Risk of Disease After Isoniazid Preventive Therapy for Mycobacterium tuberculosis Exposure in Young HIV-uninfected Children. Pediatr Infect Dis J. 2015 Nov;34(11):1218-22. doi: 10.1097/INF.0000000000000874. PMID 26252568
- [Derived] Muller J, Tanner R, Matsumiya M, Snowden MA, Landry B, Satti I, Harris SA, O'Shea MK, Stockdale L, Marsay L, Chomka A, Harrington-Kandt R, Thomas ZM, Naranbhai V, Stylianou E, Mbandi SK, Hatherill M, Hussey G, Mahomed H, Tameris M, McClain JB, Evans TG, Hanekom WA, Scriba TJ, McShane H, Fletcher HA. Cytomegalovirus infection is a risk factor for tuberculosis disease in infants. JCI Insight. 2019 Dec 5;4(23):e130090. doi: 10.1172/jci.insight.130090. PMID 31697647
- [Derived] Bunyasi EW, Tameris M, Geldenhuys H, Schmidt BM, Luabeya AK, Mulenga H, Scriba TJ, Hanekom WA, Mahomed H, McShane H, Hatherill M. Evaluation of Xpert(R) MTB/RIF Assay in Induced Sputum and Gastric Lavage Samples from Young Children with Suspected Tuberculosis from the MVA85A TB Vaccine Trial. PLoS One. 2015 Nov 10;10(11):e0141623. doi: 10.1371/journal.pone.0141623. eCollection 2015. PMID 26554383
- [Derived] Matsumiya M, Harris SA, Satti I, Stockdale L, Tanner R, O'Shea MK, Tameris M, Mahomed H, Hatherill M, Scriba TJ, Hanekom WA, McShane H, Fletcher HA. Inflammatory and myeloid-associated gene expression before and one day after infant vaccination with MVA85A correlates with induction of a T cell response. BMC Infect Dis. 2014 Jun 9;14:314. doi: 10.1186/1471-2334-14-314. PMID 24912498

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational Vaccine | Control Group
Started | 1399 | 1398
Completed | 1294 | 1303
Not Completed | 105 | 95
Not completed — Lost to Follow-up | 61 | 65
Not completed — Withdrawal by Subject | 36 | 25
Not completed — Death | 7 | 4
Not completed — Other study discontinuation | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational Vaccine | Control Group | Total
Number analyzed (Participants) | 1399 | 1398 | 2797
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1399 | 1398 | 2797
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | .401 (.039) | .399 (.037) | .400 (.038)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 691 | 682 | 1373
  Male | 708 | 716 | 1424
Region of Enrollment [Number; unit: participants]
  South Africa | 1399 | 1398 | 2797

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Safety Profile of MVA85A/AERAS-485 in Bacillus Calmette-Guerin (BCG) -Vaccinated, HIV-negative Infants.
Description: Adverse events (AE) were collected for 28 days after vaccination. The subject's parent or guardian recorded information regarding occurrences of solicited adverse events in diary cards through 7 days after vaccination. Serious adverse events (SAE) were collected from the time of study vaccine dosing throughout the entire study. A safety cohort (the first 330 infants enrolled) also had serum chemistry and hematology testing up to 28 days post-vaccination.
Time Frame: AEs recorded 28 days post-vaccination; SAEs recorded for entire study period.
Population: All subjects vaccinated.
Measure: Number (95% Confidence Interval); unit: percentage of all subjects vaccinated
Arm/Group | Investigational Vaccine | Control Group
Number analyzed (Participants) | 1399 | 1396
percentage of all subjects vaccinated | 95.9 [94.7 to 96.8] | 83.7 [81.7 to 85.6]

2. Secondary Outcome: To Evaluate the Efficacy of the MVA85A/AERAS-485 Vaccine Compared to Controls in Prevention of Tuberculosis Using an Endpoint Derived From Epidemiological Cohort Surveys in BCG Vaccinated Infants.
Description: The number (percentage) of subjects with a diagnosis of tuberculosis based on clinically-derived tuberculosis (TB) diagnostic criteria were summarized by treatment group for all subjects.
Time Frame: 15 to 36 months post-vaccination
Population: Per protocol population
Measure: Number; unit: participants with a diagnosis of TB
Arm/Group | Investigational Vaccine | Control Group
Number analyzed (Participants) | 1399 | 1395
participants with a diagnosis of TB | 32 | 39

3. Secondary Outcome: To Evaluate the Immunogenicity of the MVA85A/AERAS-485 Vaccine Compared to Controls as Described by Flow Cytometric Intracellular Cytokine Staining of CD4 and CD8 T Cells.
Description: Intracellular cytokine staining (ICS) assay immune response was expressed as the percentage of cluster of differentiation 4 (CD4) and cluster of differentiation 8 (CD8) T cells producing any one of three cytokines (IFN-γ, TNF-α, or IL-2) or any combination of the three cytokines simultaneously after stimulation with an Ag85A peptide pool on a subset of infants.
Time Frame: 28 days post-vaccination
Population: Pre-specified population subset
Measure: Median (95% Confidence Interval); unit: percentage of cytokine expressing cells
Arm/Group | Investigational Vaccine | Control Group
Number analyzed (Participants) | 27 | 27
percentage of cytokine expressing cells
  Percent cytokine expressing CD4 cells | 0.012 [0.003 to 0.038] | 0.003 [0.000 to 0.011]
  Percent cytokine expressing CD8 cells | 0.007 [0.000 to 0.011] | 0.000 [0.000 to 0.010]

4. Secondary Outcome: To Evaluate the Immunogenicity of the MVA85A/AERAS-485 Vaccine Compared to Controls as Described by the ex Vivo Enzyme Linked Immunospot (ELISPOT) Test Used in Previous MVA85A/AERAS-485 Human Trials.
Description: An ex vivo IFN-γ ELISPOT assay was used to assess specific T cell responses to an Ag85A peptide pool for a subset of infants.
Time Frame: 7 days post-vaccination
Population: Pre-specified population subset
Measure: Median (95% Confidence Interval); unit: SFC per million PBMCs
Arm/Group | Investigational Vaccine | Control Group
Number analyzed (Participants) | 27 | 27
SFC per million PBMCs | 143.000 [107.000 to 295.350] | 1.000 [0.000 to 2.000]

5. Secondary Outcome: To Evaluate the Immunogenicity of the MVA85A/AERAS-485 Vaccine Compared to Controls as Described by the University of Capetown (UCT) Whole Blood Intracellular Cytokine Assay.
Description: Frequencies of CD4 and CD8 T cells expressing cytokines (IFN-γ, IL-2 and TNF-α) following stimulation of whole blood with an Ag85A peptide pool were also measured by flow cytometry for a subset of infants.
Time Frame: 28 days post-vaccination
Population: Pre-specified population subset
Measure: Median (95% Confidence Interval); unit: percentage of cytokine expressing cells
Arm/Group | Investigational Vaccine | Control Group
Number analyzed (Participants) | 17 | 19
percentage of cytokine expressing cells
  Percent IL2/IFN-gamma/TNF expressing CD4 cells | 0.030 [0.022 to 0.079] | 0.001 [0.000 to 0.001]
  Percent IL2/IFN-gamma/ TNF expressing CD8 cells | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]

6. Secondary Outcome: To Discover Correlates of Protection From Tuberculosis in Infants Vaccinated With MVA85A/AERAS-485.
Description: Investigations for determining correlates of immune protection to TB will not be completed as planned because the study did not show TB protection in MVA85A/AERAS-485 recipients.
Time Frame: 15 to 36 months post-vaccination
Arm/Group | Investigational Vaccine | Control Group
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: To Evaluate the QuantiFERON Conversion Rate at Final Study Assessment in MVA85A/AERAS-485 Recipients Compared to Controls in Infants Without a Diagnosis of Tuberculosis During the Trial.
Description: The number (percentage) of infants with QuantiFERON conversions at any time on the study were summarized by treatment group.
Time Frame: 15 to 36 months post-vaccination
Population: Per protocol population who were quantiferon negative at baseline.
Measure: Number; unit: participants
Arm/Group | Investigational Vaccine | Control Group
Number analyzed (Participants) | 1398 | 1394
participants | 178 | 171

ADVERSE EVENTS:
Description: Two subjects within the control group were randomized but did not receive control vaccination.
Arm/Group | Investigational Vaccine | Control Group
Serious Adverse Events (participants affected / at risk) | 257/1399 | 258/1396
Other Adverse Events (participants affected / at risk) | 1319/1399 | 1064/1396
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Vaccine (N=1399) | Control Group (N=1396)
Abscess (Infections and infestations) | 1 (1) | 3 (3)
Bronchiolitis (Infections and infestations) | 10 (11) | 8 (8)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Bronchopneumonia (Infections and infestations) | 27 (29) | 28 (30)
Burn infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 2 (2)
Croup infectious (Infections and infestations) | 8 (8) | 11 (12)
Dysentery (Infections and infestations) | 1 (1) | 1 (1)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 91 (101) | 88 (94)
Hepatitis A (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 2 (2) | 2 (2)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 25 (26) | 29 (30)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Measles (Infections and infestations) | 2 (2) | 0 (0)
Meningitis (Infections and infestations) | 3 (3) | 2 (2)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Meningitis tuberculous (Infections and infestations) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 3 (3) | 2 (2)
Pneumonia (Infections and infestations) | 31 (35) | 25 (27)
Pneumonia measles (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 2 (2)
Pulmonary tuberculosis (Infections and infestations) | 6 (6) | 5 (5)
Respiratory tract infection (Infections and infestations) | 6 (6) | 10 (10)
Sepsis (Infections and infestations) | 3 (3) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 2 (2) | 3 (3)
Tuberculosis (Infections and infestations) | 5 (5) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 3 (3)
Urinary tract infection (Infections and infestations) | 8 (8) | 4 (4)
Varicella (Infections and infestations) | 1 (1) | 1 (1)
Kwashiorkor (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 2 (2) | 1 (1)
Encephalitis (Nervous system disorders) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 7 (7) | 12 (12)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal functional disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Hepatosplenomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Balanitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cryptorchism (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Sudden death (General disorders) | 1 (1) | 0 (0)
HIV test positive (Investigations) | 0 (0) | 1 (1)
Accidental drug intake by child (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Accidental exposure (Injury, poisoning and procedural complications) | 0 (0) | 3 (4)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Near drowning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumonitis chemical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 7 (7) | 10 (10)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Finger amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Vaccine (N=1399) | Control Group (N=1396)
Rhinitis (Infections and infestations) | 65 (67) | 79 (79)
Upper respiratory tract infection (Infections and infestations) | 183 (192) | 172 (180)
Hypophagia (Metabolism and nutrition disorders) | 321 (389) | 285 (357)
Insomnia (Psychiatric disorders) | 398 (513) | 359 (447)
Hypersomnia (Nervous system disorders) | 376 (478) | 324 (419)
Somnolence (Nervous system disorders) | 295 (368) | 237 (296)
Diarrhoea (Gastrointestinal disorders) | 259 (308) | 216 (245)
Vomiting (Gastrointestinal disorders) | 191 (240) | 157 (199)
Injection site erythema (General disorders) | 1121 (1183) | 446 (459)
Injection site exfoliation (General disorders) | 143 (143) | 13 (13)
Injection site pain (General disorders) | 363 (421) | 154 (175)
Injection site swelling (General disorders) | 1050 (1146) | 267 (273)
Injection site warmth (General disorders) | 473 (561) | 222 (279)
Irritability (General disorders) | 523 (659) | 431 (553)
Pyrexia (General disorders) | 372 (449) | 271 (323)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restrictions on the PI include submission of study data as an Investigator's Brochure prior to publication, sponsor's review (for a period of 60-180 days from the time submission to the sponsor for review), correction of factual errors, accommodation of reasonable comments of sponsor relating to regulatory submissions/interpretation of the Study Data (including assertion of safety and efficacy).